CLINICAL TRIAL: NCT05256576
Title: KORE-INNOVATION: a Prospective, Multi-site Clinical Trial to Implement and Analyse the Effects of an Innovative Perioperative Care Pathway to Reduce Complications for Patients with Ovarian Cancer
Acronym: KORE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Kliniken Essen-Mitte (Other)
Responsible Party: Principal Investigator, Melisa Gulhan Inci, Attending physician, Charite University, Berlin, Germany
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 01NVF18021
Record Dates: First submitted 2022-01-05; First posted 2022-02-25 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Ovary Cancer; Fallopian Tube Cancer; Peritoneum Cancer; Frailty
Keywords: Perioperative care; Prehabilitation; Enhanced Recovery after Surgery; Patient Empowerment; Postoperative Complications
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms; Frailty; Patient Participation; Postoperative Complications

STUDY DESIGN:
Intervention Model Description: multi-center, controlled, open-ended intervention study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Control Group 1 (No Intervention): Historic control group from both study sites: patients who took part in the FRAILTY study at Charité University hospital Berlin, as well as patients who were treated for OC at Evangelische Kliniken Essen Mitte during the same time period. Retrospective analysis looking at some of the main outcome variables will be conducted.
- Control Group 2 (No Intervention): Prospective control group: patients who undergo treatment for OC at both sites. Main outcomes are determined while under standard hospital care before start of the change management and implementation of the new intervention.
- Control Group 3 (No Intervention): Control group for health economical analysis to determine the cost-effectiveness of the new intervention.
- Intervention Group (Experimental): Intervention Group undergoing the new multi-modal perioperative care pathway, including the implementation of ERAS pathway, in combination with a tri-modal prehabilitation program following a comprehensive frailty assessment.
  Interventions: Other: Implementation of an innovative multi-modal peri-operative care pathway

INTERVENTIONS:
Other: Implementation of an innovative multi-modal peri-operative care pathway — The innovative multi-modal care pathway includes the implementation of the ERAS pathway, as well as the introduction of a patient-specific tri-modal prehabilitation program. This consists of a physical fitness, nutrition, and patient empowerment intervention.
  Arms: Intervention Group

SUMMARY:
KORE-INNOVATION is a multi-center clinical study aiming to implement and analyze an innovative care pathway to reduce perioperative complications for patients undergoing surgical treatment for ovarian cancer.

This is achieved by a structured, multidisciplinary implementation of the ERAS pathway, as well as introducing a tri-modal prehabilitation program, following a comprehensive frailty-assessment. The patient-individualized prehabilitation program consists of a structured plan to improve physical fitness, nutritional status, as well as patient empowerment. The aim of the study is to reduce perioperative morbidity and mortality, as well as improvement in quality of life.

DETAILED DESCRIPTION:
The treatment of patients with ovarian, fallopian tube or peritoneal cancer (OC) usually consists of a primary operation, followed by platinum-based chemotherapy and targeted maintenance therapy. According to various studies, complete macroscopic resection is considered the most important predictive factor for overall survival. Due to a lack of early detection, the majority of OC-cases are diagnosed at an advanced tumor stage. Therefore, the surgical treatment is often characterized by multi-visceral resections, in order to achieve complete macroscopic resection of the tumor mass. The rate of serious postoperative complications after debulking surgery (CDC III°-V° (Clavien-Dindo-Classification)) is about 29%. These complications are often associated with longer hospital stays and a delay in the start of the consecutive treatment, which is crucial for the overall prognosis and quality of life of OC-patients.

This study aims to implement and analyze the effect of an innovative multimodal care pathway to reduce the rate of serious complications 30 and 60 days postoperatively in patients with a primary diagnosis of OC or first platinum-sensitive recurrence of an OC, compared to patients undergoing routine treatment. The new care pathway consists of two main components: firstly, a frailty-adapted, individualized tri-modal prehabilitation program, consisting of a respective physical fitness module, an individualized nutrition plan, as well as patient empowerment. The empowerment module aims to educate patients to make informed decisions and take an active role in the recovery process, as well as build psychological resilience and activate psychosocial resources through individual and group-coaching sessions. Secondly this is combined with the implementation of the established perioperative ERAS (Enhanced Recovery after Surgery)-concept, in order to provide optimized care to patients with OC, as well as reduce the length of hospital stay and reduce health-care costs.

This study is a prospective, multicenter, controlled interventional study consisting of three phases. 1. Baseline phase, including the analysis of a prospective control group by monitoring perioperative patient care under standard care conditions. 2. Change management, which entails the preparation of the intervention phase. This consists of the integration of the new treatment procedures (prehabilitation and ERAS-pathway) into regular care. The establishment of interdisciplinary and inter-professional care teams, as well as the implementation of a training program are additional key factors. 3. Intervention phase, which entails the treatment of patients according to the new care pathway and the analysis of its effects in a prospective intervention group.

The "KORE-INNOVATION" project funded by the government and has been in the preparatory phase since July 2020.The baseline phase was conducted from April 2021 until October 2021. Change management took place from July 2021 until November 2021. The intervention phase started in December 2021 and will be going forward until June 2023.

To the best of our knowledge, this is the first attempt to implement a multimodal care pathway introducing an individualized frailty adapted, tri-modal prehabilitation program in combination with the ERAS-pathway to reduce postoperative morbidity and mortality, length of hospital stay, and health-care costs in patients with OC.

ELIGIBILITY:
Inclusion Criteria:

* Women with primary diagnosis of ovarian, fallopian tube or peritoneal cancer and primary surgical treatment (all histological subgtypes, all FIGO-stages)
* women with first recurrence of ovarian, fallopian tube or peritoneal cancer and primary surgical treatment (all histological subgtypes, all FIGO-stages)
* patients who have given and signed informed consent-forms

Exclusion Criteria:

* inoperable situs
* neoadjuvant chemotherapy
* simultaneous diagnosis of secondary primary tumors (except for breast cancer)
* dementia or other psychological diseases, that impair comprehence and compliance
* pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — eligibility is based on having been diagnosed with Ovarian cancer (OC)
Enrollment: 465 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Severe postoperative complications Clavien Dindo Classification III-V | up until postoperative day 60
  CDC III-V

SECONDARY OUTCOMES:
Postoperative complications Clavien Dindo Classification I-II | up until postoperative day 60
  CDC I-II
Postoperative morbidity | post-operative day 30, 60, 90
Length of hospital stay | up until postoperative day 90
Re-hospitalisation-rate | up until postoperative day 90
Hospital staff compliance | up until postoperative day 60
  Compliance to ERAS-items will be monitored and entered into the EIAS database for ERAS-compliance monitoring
Fried Frailty assessment modified by Inci | 3 weeks pre operation up until 30 days post operation
  A comprehensive geriatric asessment according to Fried's frailty assessment will be conducted. This includes the following tests: timed up and go test, and grip strength test. Questions included in the assessment are: weight loss >5kg in the past year, occurence of fatigue in the past week, activity level. Patients are then grouped into three categories: non-frail, pre-frail, and frail.
Postoperative mortality | up until postoperative day 90
EORTC QLQ-C30 questionnaire | up until postoperative day 60
EQ-5D-3L questionnaire | up until postoperative day 60
EORTC QLQ-OV 28 questionnaire | up until postoperative day 60
Questionnaire regarding outpatient health care expenses of patients | up until postoperative day 60

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Evangelische Kliniken Essen Mitte, Essen, North Rhine-Westphalia
  - Charité University Hospital Berlin, Berlin, State of Berlin

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Inci MG, Sehouli J, Schnura E, Lee M, Roll S, Reinhold T, Klews J, Kaufner L, Niggemann P, Groeben H, Toelkes J, Reisshauer A, Liebl M, Daehnert E, Zimmermann M, Knappe-Drzikova B, Rolker S, Nunier B, Algharably E, Pirmorady Sehouli A, Zwantleitner L, Krull A, Heitz F, Ataseven B, Chekerov R, Harter P, Schneider S. The KORE-INNOVATION trial, a prospective controlled multi-site clinical study to implement and assess the effects of an innovative peri-operative care pathway for patients with ovarian cancer: rationale, methods and trial design. Int J Gynecol Cancer. 2023 Aug 7;33(8):1304-1309. doi: 10.1136/ijgc-2023-004531. PMID 37208019